CLINICAL TRIAL: NCT04949217
Title: An Exploratory Randomized Controlled Study of Arthroscopic Inlay Bristow Procedure for Recurrent Anterior Shoulder Dislocation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2021039
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Shoulder Dislocation
Keywords: bristow; shoulder dislocation
MeSH Terms: conditions — Shoulder Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inlay Bristow Group (Experimental): Inlay Bristow procedure
  Interventions: Procedure: Inlay Bristow
- Onlay Bristow Group (Active Comparator): Onlay Bristow procedure
  Interventions: Procedure: Bristow

INTERVENTIONS:
Procedure: Inlay Bristow — A modified Bristow procedure
  Other Names: Cuistow
  Arms: Inlay Bristow Group
Procedure: Bristow — Traditional Bristow procedure
  Arms: Onlay Bristow Group

SUMMARY:
To evaluate the clinical and radiographic outcomes of arthroscopic inlay bristow procedure in treating recurrent anterior shoulder instability.

DETAILED DESCRIPTION:
Aim: To compare the clinical and radiographic outcomes following the arthroscopic Chinese Unique Inlay Bristow (Cuistow) procedure and the arthroscopic Bristow procedure.

Background: The Cuistow procedure is a modified Bristow surgery in which a Mortise and Tenon structure was added to the contact surface between the coracoid tip and the glenoid. In previous retrospective study, patients received Cuistow procedure have satisfying clinical performance and excellent postoperative bone healing rate (96.1%). However, no prospective randomized controlled trial was performed.

Methods: 70 patients with recurrent anterior shoulder instability were included and randomized to either an arthroscopic Cuistow procedure or arthroscopic Bristow procedure. Radiological evaluations with 3D CT scan were performed preoperatively, immediately after the operation, and postoperatively at three months and during the final follow-up (more than 2 years). Clinical assessment for a minimum of 24 months including the 10-point visual analog scale for pain and subjective instability, University of California at Los Angeles scoring system (UCLA score), American Shoulder and Elbow Surgeons score (ASES score), ROWE score, Subjective Shoulder Value (SSV) and active range of motion were completed by independent observers and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent anterior shoulder instability based on medical history, physical examination, and radiological results.
* A glenoid defect ≥10% but <25%
* Participation in high-demand (collision and overhead) sports combined with the presence of a glenoid defect <25% of the glenoid or without defect
* Failure after Bankart repair

Exclusion Criteria:

* Multi-directional shoulder instability
* Uncontrolled epilepsy
* History of receiving Bristow-Latarjet procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-17 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Bone union rate | 3-month postoperatily
  Bone healing was observed in 3D-CT. The bone healing rate was obtained by dividing the number of people who achieved bone healing by the total number of people
Bone union rate | 2-year postoperatively
  Bone healing was observed in 3DCT. The bone healing rate was obtained by dividing the number of people who achieved bone healing by the total number of people
ASES score | 2-year postoperatively
  The ASES score (Michener 2002) is a 10-item measure of shoulder pain and function. Pain is assessed on a 10-cm visual analog scale (VAS) and accounts for 50% of the total score. The remaining 50% of the score is determined by the responses to 10 4-point Likert-scale questions related to physical function.

SECONDARY OUTCOMES:
dislocation rate | 2-year postoperatively
  The dislocation rate was obtained by dividing the number of people who dislocated postopratively by the total number of people
VAS for pain score | 2-year postoperatively
  The visual analog scale (VAS) for pain score is the most commonly used to describe pain levels in patients, ranging from 0 to 10, with a higher score indicating more intense pain.
Active shoulder ranges of motion | 2-year postoperatively
  internal rotation at the side, and external and internal rotation at 90° of abduction

CONTACTS AND LOCATIONS:
Overall Officials: Guoqing Cui, Study Chair — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No